CLINICAL TRIAL: NCT05197959
Title: The Feasibility of rTMS and Sensorimotor Training Task for the Treatment of Complex Regional Pain Syndrome: A Pilot Study
Brief Title: Treatment of Complex Regional Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Aimee Nelson, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 777999
Record Dates: First submitted 2021-12-07; First posted 2022-01-20 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Complex Regional Pain Syndrome
Keywords: repetitive transcranial magnetic stimulation; sensorimotor training; complex regional pain syndrome
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A-Control (No Intervention): Participants in this arm will not experience any intervention during a 4 week period of time. Participants will experience their standard medical care.
- Group B-rTMS and sensorimotor training (Experimental): Repetitive transcranial magnetic stimulation (rTMS) will be delivered at 10 Hz, 2000 pulses targeting the hand representation of the left primary motor cortex. Immediately following rTMS, participants will perform sensorimotor training. Nerve stimulation will be applied to the second through fifth digits and the wrist of the affected limb to cue movement. This intervention will be performed approximately 4 days per week for 4 weeks. In addition, participants will experience their standard medical care.
  Interventions: Device: Repetitive transcranial magnetic stimulation; Other: Sensorimotor training
- Group C-Sensorimotor training (Experimental): Participants will perform sensorimotor training intervention. Nerve stimulation will be applied to the second through fifth digits and the wrist of the affected limb to cue movement. This intervention will be performed approximately 4 days per week for 4 weeks. In addition, participants will experience their standard medical care.
  Interventions: Other: Sensorimotor training

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive, non-painful procedure used to relieve chronic pain and promote short-term changes. The abductor pollicis brevis (APB) muscle of the left motor cortex will be targeted using neuronavigation software. 2000 pulses will be delivered at 10 Hz stimulation. Stimulation will be delivered at 80% of the resting motor threshold obtained from the right APB muscle. The delivery of rTMS requires ~ 11.5 minutes in total.
  Other Names: rTMS; Repetitive TMS
  Arms: Group B-rTMS and sensorimotor training
Other: Sensorimotor training — Sensorimotor training is a non-invasive, non-painful procedure using nerve stimulation to cue motor action. Nerve stimulation is applied the second through the fifth digit and the median nerve at the wrist. This stimulation is used to cue a motor action. The number of stimulations will indicate the amount of movements. For example, two pulses of stimulations to the index finger would require two flexion and extension actions with the index finger. Once the stimulation occurs, the participant will flex and extend the corresponding area where the nerve stimulation was felt. This will take ~ 30 minutes to complete.
  Arms: Group B-rTMS and sensorimotor training; Group C-Sensorimotor training

SUMMARY:
This study will investigate the feasibility of using repetitive transcranial magnetic stimulation (rTMS) and a sensorimotor training task to treat symptoms of pain in patients with complex regional pain syndrome (CRPS). rTMS is a non-invasive technique that involves delivering magnetic pulses in rapid succession over the area of the brain that controls movement. The sensorimotor training task involves non-invasive nerve stimulation used to cue a participant to complete motor actions. The purpose of this study is to determine whether recruitment is feasible in this patient population and patients maintain adherence to the intervention. In addition, the investigators want to determine whether rTMS combined with sensorimotor training is an effective intervention to alleviate symptoms of pain in patients with CRPS.

DETAILED DESCRIPTION:
Background: Complex regional pain syndrome (CRPS) is a chronic pain condition characterized by a constellation of sensory, motor and autonomic dysfunction (Gierthmühlen et al., 2014). CRPS can be a debilitating disorder that drastically impacts quality of life. There are two types of CRPS; type 1 in which there is no identifiable nerve injury but occurs after a known noxious event and commonly involves immobilization, and type 2 in which there is a distinct nerve injury. There are challenges in the diagnosis of CRPS and presently the Budapest criteria are modified for the relevant context of research or practice. For this study the investigators plan to use the Budapest modified research criteria as suggested (Harden et al., 2013). CRPS differs from other chronic pain conditions; neuropathic-such as radicular pain or postherpetic neuralgia, or generalized non-specific pain conditions-such as fibromyalgia; in that, pain is associated with obvious and distinct alterations in sensory processing, sympathetic nervous involvement, and motor dysfunction. Limited treatment options for these individuals currently exist, and guidelines are based on expert consensus (Goebel et al, 2019). Existing knowledge suggests that continued physiotherapy with supportive pain control and psychological treatment is the most important strategy to manage CRPS (Goebel et al, 2019).

Repetitive transcranial magnetic stimulation (rTMS) offers a potential opportunity to noninvasively treat pain in patients with CRPS. Some studies have illustrated the analgesic effects of rTMS in patients with CRPS. Gaertner et al. (2018) delivered 10 Hz stimulation to the motor cortex in patients with CRPS. Patients were able to choose between one (n= 6) or five (n= 15) sessions of treatment. A significant reduction in pain was demonstrated in both groups one week following the last treatment session. There were no group differences in changes in pain. Two patients from each group maintained a >50% reduction in pain relief beyond 6 weeks post treatment. Further, Piceralli et al. (2010) observed a reduction in pain following 10 sessions of 10 Hz rTMS applied to the motor cortex in a group of 12 patients with CRPS. Additionally, Pleger et al. (2004) found that one session of rTMS applied to the motor cortex was sufficient to cause pain relief, however the duration of relief was experienced for only 45 minutes after stimulation. rTMS has been also used in other chronic pain conditions such as neuropathic pain (NP). Sham controlled studies have demonstrated the analgesic effects of rTMS applied to the primary motor cortex on NP symptoms in patients with spinal cord injury (Defrin et al., 2007; Jette et al., 2013; Yilmaz et al., 2014; Sun et al., 2019). These latter effects occur immediately following treatment (Jette et al., 2013) and persist up to six-weeks post-treatment (Yilmaz et al., 2014).

Although the chronic pain condition may vary, analgesic effects of rTMS are suggested to be a result of modulation of nociceptive inhibitory circuits from stimulation of the motor cortex (Lefaucheur et al., 2008; Nizard et al., 2012). This stimulation may cause changes in glutamatergic or GABAergic neurotransmitter pathways leading to a suppression of pain sensation (Lefaucheur et al., 2008; Ciampi De Andrade et al., 2014). Additionally, rTMS facilities neuroplasticity and the retraining of cortical circuits. This can be used to restore cortical activity that is altered in patients with CRPS (León et al., 2018).

Unlike other chronic pain conditions, the aim of CRPS treatment includes halting the progression of the disease early and thereby decreasing pain, rather than targeting pain alone. One approach is to reinforce afferent connections between the affected limb and the somatosensory cortex. In addition to pain, CRPS is associated with structural and functional changes of the somatosensory, primary motor, and supplementary motor areas (Urits et al., 2018; Echalier et al., 2020). Specifically, cortical representations of the affected limb in the somatosensory cortex are smaller and possess greater overlap with adjacent areas (Swart et al., 2009; Pietro et al., 2013). This is speculated to be a result of a decrease in afferent input originating from the periphery (Legrain et al., 2011; Moseley et al., 2012). Additionally, this reorganization is reinforced by the minimal usage of the affected limb by patients in order to avoid pain (Echalier et al., 2020). As such, this begins to raise the question, as to whether a sensorimotor task that stimulates afferent input originating from the periphery may aid in reinstating somatosensory cortical territory and ultimately aid in pain relief in these patients.

The objective of this study is to investigate the feasibility of the study procedures in a feasibility study involving 18 patients. In addition, the use of rTMS paired with a sensorimotor training task will be investigated in CRPS I patients, to induce positive neuroplastic changes so as to effect temporary and long-term pain relief. rTMS will be delivered to the primary motor cortex controlling the hand to create an environment within the sensory motor cortex that promotes neuroplasticity. This is accomplished through high frequency rTMS which increases cortical excitability (León et al., 2018). This in turn promotes intraneuronal connectivity and reorganization achieved through sensorimotor integration provided by the sensorimotor training task. In this task, digits two through five and the wrist on the affected hand will be non-invasively stimulated individually and require the participant to make a movement with that digit or wrist.

Study design: All participants will provide written informed consent. The patients will maintain their current medications and physiotherapy throughout the duration of the experiment. Participants will be randomly allocated into one of three groups. All groups will continue to have conservative care and physiotherapy as appropriate to their condition. Group A-control will not experience the intervention, group B will experience the rTMS and sensorimotor training intervention. Group C will experience the sensorimotor training intervention only. The intervention will be performed approximately 4 days per week for 4 weeks. During this 4 week time period, participants in group A will not experience any intervention.

Study intervention procedure: Repetitive transcranial magnetic stimulation (rTMS) will be applied to the left motor cortex representation of the right abductor pollicis brevis (APB) muscle regardless of affected hand (Sun et al., 2019). Surface electromyography (EMG) electrodes will be placed on the skin overlying the APB muscle. The skin site will be cleaned using alcohol prior to adhering the disposable electrodes. Next the location of the right APB muscle in the left hemisphere will be determined by delivering stimuli at ~50 % maximum stimulator output (MSO) over the approximate location of the right APB representation and adjusting the coil position until large and consistent motor evoked potentials (MEPs) are elicited. If the investigators are unable to get a MEP from the APB muscle, the investigators will attempt to obtain the MEP from the first dorsal interosseous muscle. The spatial position that elicits large and consistent MEP's will be recorded using Brainsight Neuronavigation. This location is referred to as the motor hotspot and will be used throughout the intervention. This procedure will take ~15min to complete. rTMS stimulation will be applied to the identified motor hotspot at 80% resting motor threshold (RMT) (Sun et al., 2019). RMT will be performed each time rTMS is delivered and at T0, T1 and T2. To obtain RMT, the patient will receive single pulses of TMS to the APB hotspot. The RMT is defined as the minimum TMS intensity that evokes a motor response of 50 μV in 5 out of 10 consecutive trials when the APB muscle is at rest. This procedure will take ~5min to complete. Following calibration of the RMT, the patient will receive the rTMS stimulation using a 90 mm figure-8 coil. The coil will be positioned tangent with the scalp at 45° from midline, and the handle of coil will be pointed 5° backward and laterally. The patient will receive 2000 pulses at 10 Hz stimulation frequency (Sun et al., 2019; Yilmaz et al., 2014; Jette et al., 2013; Kang et al., 2009; Nardone et al., 2017). One hundred and sixty-seven trains will be delivered for a duration of 1.2s (3s inter-train interval) (Sun et al., 2019). rTMS delivery will require ~11.5 min to complete.

For participants in Group B, immediately following rTMS the participant will engage in a sensorimotor training task that involves digital and median nerve stimulation applied to each individual digit separately using ring electrodes and the median nerve using a bar electrode. Participants in group C will experience the sensorimotor training task without rTMS before hand. During the sensorimotor training task participants will experience nerve stimulation to either one of their digits (2-5) or the median nerve at the wrist. A trial will commence when one of the areas (digit or wrist) is stimulated for 2 ms with either one or two pulses of stimulation. The number of stimulations will indicate the amount of movements. For example, two pulses of stimulations to the index finger would require two flexion and extension actions. Once the stimulation occurs, the participant will flex and extend the corresponding area where the nerve stimulation was felt. This training will require approximately 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of CRPS type 1 affecting one of their hands

Exclusion Criteria:

* A known history of moderate to severe chronic pain in other parts of the body
* Daily use of opioids prior to the CRPS diagnosis
* Contraindications to transcranial magnetic stimulation
* Known psychological diagnosis affecting comprehension
* Inability to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Ability to recruit 6 patients in each group over a 6-month period | Immediately following the 4 week intervention.
  Ability to recruit 6 patients in each group over a 6-month period at the chronic pain clinic at St Joseph's Healthcare Hamilton.
Compliance of treatment sessions as proposed | Immediately following the 4 week intervention.
  Percentage of participants that completed all treatment sessions. We expect >90% patients in each group to adhere to sessions.

SECONDARY OUTCOMES:
Complex Regional Pain Syndrome Severity Scale | 1 week before intervention, immediately before intervention, immediately following intervention, 6 months after intervention
  Questionnaire used to assess the severity of CRPS using 17 clinically assessed signs/symptoms of CRPS. The questions are divided into self reported symptoms and signs observed on examination. Results are reported as percent yes from 0 to 100 percent. Higher score means worse outcome.
PROMIS-29 v2.0 Profile | 1 week before intervention, immediately before intervention, immediately following intervention, 6 months after intervention
  Using numerical rating (0 to 5) to assess seven health domains including physical function, anxiety, depression, fatigue, sleep disturbances, ability to participate in social roles and activities, and pain interference. Each category consists of 4 questions. Also uses a numerical rating to asses pain intensity (0-10).
Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) Pain Score | 1 week before intervention, immediately before intervention, immediately following intervention, 6 months after intervention
  A seven item questionnaire based on bedside sensory tests used to identify pain of neuropathic origin from nociceptive pain. Five questions are used to understand characteristics of pain and two questions require rubbing and pressing on the painful area to determine the pain response. Scored from 0 to 24. A score of 12 or greater suggests pain of predominantly neuropathic origin.
The Rainbow Pain Scale | 1 week before intervention, immediately before intervention, immediately following intervention, 6 months after intervention
  Used to measure the severity of allodynia type pain using sensory assessments of the affected limb. Seven different sized monofilaments (von Frey filaments) are applied at different force levels to the painful area. The size of the monofilament and force of application increases until the participant has indicated that the stimulus has become painful and the corresponding rainbow pain scale category is recorded. Recorded as force level from 0.04 g to 15 g and monofilament size from 2.55 to 5.18 that elicited a painful response. Lower force and size values means worse outcome.
Douleur Neuropathique 4 (DN4 Scale) | 1 week before intervention, immediately before intervention, immediately following intervention, 6 months after intervention
  A 10 item questionnaire used to determine the probability that the pain is neuropathic in origin. Each question consist of either a yes or no answer and the number of yes answers are totalled between 0 to 10. Higher score means worse outcome.
Medication Use | 1 week before intervention, immediately before intervention, immediately following intervention, 6 months after intervention
  Quantity of daily narcotics or non-narcotics used.
Patient Perceived Global Index of Change (PGIC) | 1 week before intervention, immediately before intervention, immediately following intervention, 6 months after intervention
  1-7 Likert Scale: Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse.
Assessments of swelling and skin discolouration using pictures and videos | 1 week before intervention, immediately before intervention, immediately following intervention, 6 months after intervention
  Pictures and videos of the affected hand and wrist will be taken in different postures including: supination-pronation; flexion-extension of wrist, abduction-adduction of wrist; flexion-extension movements of fingers.These pictures will be used to assess physical symptoms of CRPS including swelling and skin discolouration.
The Patient Rated Wrist/Hand Evaluation (PRWHE scale) | 1 week before intervention, immediately before intervention, immediately following intervention, 6 months after intervention
  A 15 item questionnaire used to measure pain in the wrist and its affect on activities of daily living. Questions are split into 3 categories consisting of the amount of pain in the wrist during different actions, difficulty in completing activities of daily living, and difficulties in completing activities of daily living before the injury occurred. Sum of function and pain scores is reported from 0 to 100. Higher score means worse outcome.
Sensory nerve action potentials | 1 week before intervention, immediately before intervention, immediately following intervention, 6 months after intervention
  Will be obtained through digital nerve, median nerve, and ulnar nerve stimulation of the affected and non-affected hand. Sensory nerve action potentials will be recorded using removable adhesive EMG electrodes positioned over the medial elbow and wrist.
Somatosensory evoked potentials | 1 week before intervention, immediately before intervention, immediately following intervention, 6 months after intervention
  Will be obtained through stimulation of the digital nerve for each digit, alongside the median and ulnar nerves of the affected and non-affected hand. Somatosensory evoked potentials will be recorded at the somatosensory cortex contralateral to the stimulated hand.
Hoffman reflex | 1 week before intervention, immediately before intervention, immediately following intervention, 6 months after intervention
  Will be obtained by stimulating the median nerve at the wrist using a bar electrode. Muscle activity will be recorded using EMG activity in the APB muscle while the participant maintains 5% of maximum voluntary contraction (MVC).
Von Frey Filaments | 1 week before intervention, immediately before intervention, immediately following intervention, 6 months after intervention
  Von Frey Filaments are used to measure mechanical sensitivity on the hand. Monofilaments are applied to the hand in decreasing diameter until the application can no longer be felt. This represents the mechanical sensitivity of the tested area to tactile perception.
Johnson Vanboven Phillips Domes (JVP) | 1 week before intervention, immediately before intervention, immediately following intervention, 6 months after intervention
  Used to measure spatial acuity on the hand. Domes of decreasing grading are applied to the hand. Grading is used to represent the distances between ridges on the dome. The domes are applied until the dome with the finest grating that is correctly identified 75 percent of the time is found. This represents the spatial acuity limit of the tested area.
Brain derived neurotrophic factor (BDNF) | Immediately before intervention, immediately following intervention
  BDNF will be used as a measure of neuroplasticity. Blood will be drawn from 12-h fasted participants in the morning. A 10-ml increased silica act clot activator, silicone-coated tube (red top) will be used. Blood collected in the red top tube will be allowed to clot by leaving it undisturbed at room temperature for approximately 45 minutes and then centrifuged at 2,000 x g for 10 minutes at 4 °C. Serum will be pipetted into a fresh tube, aliquoted and stored at -80 °C prior to use. Protein levels of BDNF and NGF will be measured in serum using enzyme-linked immunosorbent assays (ELISAs).
Nerve growth factor (NGF) | Immediately before intervention, immediately following intervention
  NGF will be used as a measure of neuroplasticity and pain. Blood will be drawn from 12-h fasted participants in the morning. A 10-ml increased silica act clot activator, silicone-coated tube (red top) will be used (This will be the same tube used for BDNF). Blood collected in the red top tube will be allowed to clot by leaving it undisturbed at room temperature for approximately 45 minutes and then centrifuged at 2,000 x g for 10 minutes at 4 °C. Serum will be pipetted into a fresh tube, aliquoted and stored at -80 °C prior to use. Protein levels of BDNF and NGF will be measured in serum using enzyme-linked immunosorbent assays (ELISAs).

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton King Campus, Hamilton, Ontario, Canada